CLINICAL TRIAL: NCT00041106
Title: Phase II Study Of Cisplatin, Gemcitabine, And ZD 1839 (IRESSA) (IND #61187; NSC 715055) For The Treatment Of Advanced Urothelial Tract Carcinoma
Brief Title: Gefitinib Plus Combination Chemotherapy in Treating Patients With Locally Advanced or Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02818; CALGB-90102; CDR0000069443; U10CA031946 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter
MeSH Terms: interventions — Gemcitabine; Cisplatin; Gefitinib

ARMS (1):
- Treatment (gemcitabine, cisplatin, and gefitinib) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 1 hour on day 1. Patients also receive gefitinib PO QD beginning on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete remission, partial remission, or maintain stable disease continue gefitinib PO QD for 5 years or until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: gemcitabine hydrochloride; Drug: cisplatin; Drug: gefitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: gefitinib — Given PO
  Other Names: Iressa; ZD 1839
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of the tumor. Combining chemotherapy with gefitinib may kill more tumor cells. Phase II trial to study the effectiveness of combining chemotherapy with gefitinib in treating patients who have metastatic transitional cell cancer of the urothelium

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the overall response proportion in patients with advanced carcinoma of the urothelial tract treated with cisplatin, gemcitabine (gemcitabine hydrochloride) and ZD1839 (gefitinib), given on a 21 day schedule, followed by maintenance ZD1839.

SECONDARY OBJECTIVES:

I. To describe the time to progression, progression-free survival, and overall survival in patients with advanced carcinoma of the urothelial tract treated with cisplatin, gemcitabine and ZD1839, given on a 21 day schedule, followed by maintenance ZD1839.

II. To evaluate the effect of epidermal growth factor receptor (EGFR) expression level on overall response rate and progression-free survival in patients with advanced carcinoma of the urothelial tract treated with cisplatin, gemcitabine and ZD1839, given on a 21 day schedule, followed by maintenance ZD1839.

III. To assess the toxicity of the combination of cisplatin, gemcitabine and ZD1839 given on a 21 day schedule, followed by maintenance ZD1839 in patients with advanced carcinoma of the urothelial tract.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine intravenously (IV) over 30 minutes on days 1 and 8 and cisplatin IV over 1 hour on day 1. Patients also receive gefitinib orally (PO) once daily (QD) beginning on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete remission, partial remission, or maintain stable disease continue gefitinib PO QD for 5 years or until disease progression or unacceptable toxicity occurs.

Patients are followed at least every 3 months for 1 year and then at least every 6 months until disease progression or relapse.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven transitional cell carcinoma of the urothelial tract (bladder, ureter, renal pelvis or urethra); histologic documentation of metastatic/recurrent disease is not required; clinical, but not pathologic staging, is required
* Metastatic (N2, N3 or M1) urothelial tract carcinoma; patients must not be candidates for potentially curative surgery or radiation therapy
* Patients must have measurable disease as defined below:

  * Measurable disease: lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; the bladder is not a site of measurable disease
  * Non-measurable disease: all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions; lesions that are considered non-measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Prior treatment:

  * No prior systemic chemotherapy except single-agent chemotherapy used as a radiosensitization agent; prior intravesical chemotherapy is permissible; prior adjuvant or neoadjuvant chemotherapy is not permissible
  * No prior systemic therapy for advanced urothelial carcinoma including investigational therapies such as, but not limited to, agents targeting the HER2/neu, signal transduction (including EGFR), angiogenic, immune, and cell cycle pathways
  * No prior treatment with ZD1839
  * > 4 weeks and fully recovered from major surgery, radiation, or intravesical chemotherapy
* Tumor tissue from the primary tumor or from biopsy of a metastatic site must be available for EGFR expression determination; when tissue specimens from both primary and metastatic sites are available, both must be submitted for EGFR testing; expression of EGFR is not required
* No cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers within 7 days prior to starting protocol therapy and while on protocol treatment; CYP3A4 inducers include phenytoin, carbamazepine, barbiturates, rifampin, St John's Wort, dexamethasone, modafinil, and rifapentine; single doses of dexamethasone used as an antiemetic are permitted
* No evidence of brain metastases
* Patient must have no evidence of:

  * > grade 1 pre-existing sensory or motor neuropathy
  * Active severe chronic gastrointestinal disorders including liver disease, diarrheal or emetic disorders, or malabsorptive conditions causing nausea or diarrhea
  * Active severe chronic desquamative cutaneous disorder
  * Active severe corneal disease or inflammatory ocular disorder
* No "currently active" second malignancy other than non-melanoma skin cancers; patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse
* No patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No human immunodeficiency virus (HIV) disease
* Common Toxicity Criteria (CTC) (Eastern Cooperative Oncology Group [ECOG]) performance status 0-2
* Granulocytes >= 1,500/ul
* Platelet count >= 100,000/ul
* Bilirubin =< 1.25 x upper limits of normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.0 x upper limits of normal
* Calculated creatinine clearance >= 50 ml/min

Exclusion Criteria:

* Patients must not be pregnant or engaged in nursing; men and women of reproductive age must agree to practice effective contraception in order to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-05; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria and defined as either a complete or partial response | Up to 7 years
  Exact 95% confidence intervals based on the binomial distribution will be computed.

SECONDARY OUTCOMES:
Toxicity rates assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 7 years
  Exact 95% confidence intervals based on the binomial distribution will be computed.
Progression-free survival (PFS) | From the date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 7 years
  The Kaplan-Meier product limit method will be used to estimate the PFS.
Overall survival (OS) | From the date of initiation of treatment to date of death due to any cause, assessed up to 7 years
  The Kaplan-Meier product limit method will be used to estimate the OS.

CONTACTS AND LOCATIONS:
Overall Officials: George Philips, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States